CLINICAL TRIAL: NCT01846741
Title: VNS Therapy Automatic Magnet Mode Outcomes Study in Epilepsy Patients Exhibiting Ictal Tachycardia
Brief Title: VNS Therapy Automatic Magnet Mode Outcomes Study in Epilepsy Patients Exhibiting Ictal Tachycardia (E-37)
Acronym: E-37
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epilepsy (E)-37
Record Dates: First submitted 2013-04-15; First posted 2013-05-03 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Epilepsy
Keywords: Automatic Magnet Mode (AMM); Vagus Nerve Stimulation (VNS)
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Model 106 VNS Therapy System (Other)
  Interventions: Device: M106 VNS Therapy System

INTERVENTIONS:
Device: M106 VNS Therapy System

SUMMARY:
Obtain baseline clinical outcome data (Stage 1) upon which to base a subsequent study (Stage 2) of the Model 106 VNS implantable pulse generator

DETAILED DESCRIPTION:
Prospective, observational, un-blinded, multi-site study designed to collect data on patients implanted with a Model 106 VNS Therapy System from baseline through an EMU stay of up to 5 days, and 6-month follow-up. After the 6-month follow-up, patients will continue follow-up for safety for approximately two years or until final regulatory approval of the product.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of medically refractory epilepsy with partial onset seizures suitable for implantation with the VNS Therapy System.
* Patients willing to undergo an EMU evaluation for a period of at least three days with activation of the AMM feature during that time.
* Patients must be at least 12 years old.
* Patients must be in good general health and ambulatory.
* Patient or guardian must be willing and able to complete informed consent/assent.

Exclusion Criteria:

* Patients have had a bilateral or left cervical vagotomy.
* Patients currently using, or are expected to use, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy.
* A VNS Therapy System implant would (in the investigator's judgment) pose an unacceptable surgical or medical risk for the patient.
* Patients expected to require full body magnetic resonance imaging (MRI).
* Patients have a history of implantation of the VNS Therapy.
* Patients with an IQ known or estimated to be < 70, history of depression requiring hospitalization, or suicidality as defined by DSM IV-TR that in the investigator's judgment would pose an unacceptable risk for the patient or prevent the patient's successful completion of the study.
* Patients with a history of status epilepticus within 1 year of study enrollment.
* Patients with known clinically meaningful cardiovascular arrhythmias as well as patients with clinically meaningful cardiovascular arrhythmias determined by a 24-hour Holter recording obtained during the baseline period.
* Patients dependent on alcohol or narcotic drugs as defined by DSM IV-TR within the past 2 years.
* Patients with a history of psychogenic non-epileptic seizures.
* Women who are pregnant. Women of childbearing age must take a pregnancy test and agree to use an approved method of contraception during the study.
* Patients currently enrolled in another investigational study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Begnaud, Study Director — Cyberonics, Inc.; Robert Fisher, MD, PhD, Principal Investigator — Stanford University
Locations (15):
- United States (15):
  - Phoenix, Arizona
  - Stanford, California
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Ann Arbor, Michigan
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Albany, New York
  - Durham, North Carolina
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were at least 12 years old, good general health suitable for VNS implant with refractory (drug-resistant) partial onset seizures and a history of ictal tachycardia, defined as heart rate above 100 beats per minute (bpm) during a seizure and at least a 55% increase or 35 bpm increase from baseline.
Pre-assignment Details: A total of (22) subjects were screened; (2) did not meet study criteria, (20) were treated/implanted with the AspireSR® VNS Therapy® System.
Groups:
- VNS Therapy - ITT Population: Subjects who were implanted with the AspireSR® VNS Therapy® System.
  The intent-to-treat (ITT) population is defined as all subjects with the VNS Therapy system implanted and the device had been turned on.
Period: Baseline Visit
Arm/Group | VNS Therapy - ITT Population
Started | 22
Completed | 20
Not Completed | 2
Not completed — Subject did not meet entry criteria | 2
Period: Implantation to 18-Month/End of Study
Arm/Group | VNS Therapy - ITT Population
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects implanted with VNS Therapy system
Groups:
- VNS Therapy (ITT Population): Subjects who were implanted with the AspireSR® VNS Therapy® System.
Arm/Group | VNS Therapy (ITT Population)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.6 (14.1)
Age, Customized [Median (Full Range); unit: years] | 31 [21 to 69]
Age, Customized [Number; unit: years]
  18-29 years | 9
  30-39 years | 5
  40-49 years | 2
  50-59 years | 2
  60 years or older | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 15
  Black or African American | 2
  Hispanic or Latino | 3
Cognitive Status [Number; unit: participants]
  Normal | 14
  Minimal Impairment | 6
Time from diagnosis to VNS therapy [Mean (Standard Deviation); unit: years] | 21.2 (15.3)
Time from diagnosis to VNS therapy [Median (Full Range); unit: years] | 17 [1 to 52]
Previous brain or Epilepsy surgery [Number; unit: participants]
  No | 12
  Yes | 8
Etiology [Number; unit: participants]
  Idiopathic Partial | 8
  Symptomatic Partial | 10
  Cryptogenic | 2
Family history of seizures [Number; unit: participants]
  No | 12
  Yes | 8
Seizures with auras in past 2 months [Number; unit: participants]
  No | 7
  Yes | 13

OUTCOME MEASURES:

1. Secondary Outcome: Summary of Seizures Reported by Investigators and Triple Review
Description: Seizure events were recorded during the EMU stay (only Automatic Stimulation Mode aka AutoStim ON) using vEEG and ECG to evaluate tachycardia detection algorithm performance. The threshold for the AutoStim feature (20-70%) was programmed for each subject, based upon the historical ictal elevation in heart rate for that subject, requiring the corresponding heart rate elevation above that of a moving baseline window.
  Number of seizures observed and reported by investigators during the EMU stay (several subjects had more than one type of seizure) were collected and also reviewed by three (3) independent and blinded reviewers for confirmation. Additionally, the reviewers identified new seizures while reviewing the study EMU stay vEEG.
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: ITT Population: Consists of all patients in the safety population who have any EMU performance recorded data and experienced any seizures.
Measure: Number; unit: Number of Seizures
Groups:
- Reported By Investigators: All Seizures Identified (During EMU)
- Reported by Triple Review: EMU Seizures Identified Post EMU
- Total: Seizures Reported by Investigators and Triple Reviewers
Arm/Group | Reported By Investigators | Reported by Triple Review | Total
Number analyzed (Participants) | 16 | 16 | 16
Number of Seizures
  All Seizure Types | 84 | 5 | 89
  Total Partial Seizures | 76 | 0 | 76
  Simple Partial | 37 | 0 | 37
  Complex Partial | 38 | 0 | 38
  Secondarily Generalized | 1 | 0 | 1
  Sub-Clinical | 8 | 1 | 9
  Unclassified | 0 | 4 | 4

2. Secondary Outcome: Assess Performance of the Tachycardia Detection Algorithm (Sensitivity) During an EMU Stay Based on ITT Population-Observed
Description: Sensitivity is defined as the total number of seizures detected divided by the total number of seizures during the EMU stay. Data used to support sensitivity analyses included digital ECG/EEG files, corresponding M106 device downloads, and CRF data. Seizure and non-seizure EEG segments were provided to independent reviewers to confirm seizure occurrence and define electrographic seizure onset times. Seizure onset times were then compared with observed M106 device detections at the least sensitive setting capable of detecting the seizure based on the corresponding change in heart rate. Threshold for AutoStim setting (1;70%, 2;60%, 3;50%, 4;40%, 5;30% and 6;20%). No subjects were assigned to settings 3 and 6 that had seizures with a corresponding heart rate increase of >= 50% and >= 20%, respectively. Number of participants is total number of subjects who experienced seizures during the EMU stay.
  Bootstrap confidence intervals using 3000 bootstrap samples.
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: ITT Population (Investigator Reported Seizures + Triple Review). N= represents total number of seizures.
Measure: Number (95% Confidence Interval); unit: Percent of True Positive Seizures
Groups:
- % Sensitivity: Based on Heart rate Increase Associated with Seizures by Threshold for AutoStim
Arm/Group | % Sensitivity
Number analyzed (Participants) | 16
Percent of True Positive Seizures
  >= 70% heart rate increase at Setting 1 (n=1) | 0 [NA to NA] — Confidence interval was not calculated where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated)
  >= 60% heart rate increase at Setting 2 (n=9) | 100 [NA to NA] — Confidence interval was not calculated where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated)
  >= 40% heart rate increase at Setting 4 (n=1) | 100 [NA to NA] — Confidence interval was not calculated where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated)
  >= 30% heart rate increase at Setting 5 (n=2) | 50 [NA to NA] — Confidence interval was not calculated where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated)

3. Secondary Outcome: Assess Performance of the Tachycardia Detection Algorithm (Sensitivity) During an EMU Stay Based on ITT Population-Modeled
Description: Sensitivity is defined as the total number of seizures detected divided by the total number of seizures during the EMU stay. Data used to support sensitivity analyses included digital ECG/EEG files, corresponding M106 device downloads, and CRF data. Seizure onset times were compared with modeled M106 device detections at the least sensitive setting capable of detecting the seizure based on the corresponding change in heart rate. The participants' surface ECG data collected during the trial and passed through DMSDAT, a validated bench-top simulant of the Automatic Stimulation feature, was used to produce modeled results for each threshold for AutoStim setting (1;70%, 2;60%, 3;50%, 4;40%, 5;30% and 6;20%). Number of participants is total number of subjects who experienced seizures during the EMU stay.
  Bootstrap confidence intervals using 3000 bootstrap samples.
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: ITT Population (Investigator Reported Seizures + Triple Review). N= represents total number of seizures.
Measure: Number (95% Confidence Interval); unit: Percent of True Positive Seizures
Arm/Group | % Sensitivity
Number analyzed (Participants) | 16
Percent of True Positive Seizures
  >= 70% heart rate increase at Setting 1 (n=8) | 87.5 [77 to 100]
  >= 60% heart rate increase at Setting 2 (n=12) | 100 [NA to NA] — Confidence interval was not calculated where the mean sensitivity equals to 100%
  >= 50% heart rate increase at Setting 3 (n=20) | 95 [91 to 100]
  >= 40% heart rate increase at Setting 4 (n=23) | 100 [NA to NA] — Confidence interval was not calculated where the mean sensitivity equals to 100%
  >= 30% heart rate increase at Setting 5 (n=31) | 100 [NA to NA] — Confidence interval was not calculated where the mean sensitivity equals to 100%
  >= 20% heart rate increase at Setting 6 (n=38) | 100 [NA to NA] — Confidence interval was not calculated where the mean sensitivity equals to 100%

4. Secondary Outcome: Assess Non-seizure Related Stimulation Rate Per Hour During EMU Stay and Stair Stepper Exercise Periods
Description: Each day in the EMU, subjects exercised for up to 3 minutes stepping up and down at a submaximal effort level on a step stool. Subject's resting heart rate was compared with the calculated 85% of the patient's age-predicted maximum heart rate. This calculated heart rate was then used as termination criteria for the step test.
  Non-Seizure Detection Rate (previously known as Potential False Positive Rate) is defined as the total number of non-seizure detections summed for the group divided by the total evaluable monitoring time during the EMU. The non-seizure detection rate per hour was calculated at the various tachycardia detection settings for all subjects during EMU and during exercise activities (stair stepper).
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: ITT Population. 5 participants analyzed for >=70%, 4 for >=60% setting, 8 for >=50% setting, 2 for >=40% setting, 1 for the >=30% setting.
Measure: Number (95% Confidence Interval); unit: detections per hour
Groups:
- During EMU Stay; During EMU Stay Stair-Stepper Exercise: Non-Seizure Related Stimulation Rate (AutoStim Per Hour)
Arm/Group | During EMU Stay | During EMU Stay Stair-Stepper Exercise
Number analyzed (Participants) | 20 | 20
detections per hour
  >=70%, n=5 | 0.4 [0.1 to 1.0] | 1.6 [0 to 6.4]
  >=60%, n=4 | 0.8 [0.3 to 1.4] | 4.0 [0 to 9.9]
  >=50%, n=8 | 1.2 [0.8 to 1.6] | 6.2 [2.0 to 12.2]
  >=40%, n=2 | 0.6 [NA to NA] — Confidence intervals were not calculated where number of subjects within the setting is less than or equal to 2 (acceleration can not be calculated) | 6.6 [NA to NA] — Confidence intervals were not calculated where number of subjects within the setting is less than or equal to 2 (acceleration can not be calculated)
  >= 30%, n=1 | 4.6 [NA to NA] — Confidence intervals were not calculated where number of subjects within the setting is less than or equal to 2 (acceleration can not be calculated) | 5.0 [NA to NA] — Confidence intervals were not calculated where number of subjects within the setting is less than or equal to 2 (acceleration can not be calculated)

5. Secondary Outcome: Assess Characterization of Seizures (Duration and Cessation)
Description: Clinical outcomes including seizure duration and cessation were assessed with vEEG during EMU stay. Number of seizures treated with Automatic Stimulation during EMU were evaluated. Of these seizures, those ending during the 60 second course of Automatic Stimulation were assessed and tabulated by seizure type.
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: ITT Population
Measure: Number; unit: Percent of Seizures Ended During Stim
Units Other Than Participants: Seizures Treated
Groups:
- Overall Seizures; Complex Partial Seizures; Secondary Generalized Seizures; Simple Partial Seizures; Sub-Clinical Seizures; Unknown Seizures: During AutoStim Course in The EMU
Arm/Group | Overall Seizures | Complex Partial Seizures | Secondary Generalized Seizures | Simple Partial Seizures | Sub-Clinical Seizures | Unknown Seizures
Number analyzed (Participants) | 12 | 7 | 1 | 6 | 1 | 2
Number analyzed (Seizures Treated) | 31 | 12 | 1 | 12 | 4 | 2
Percent of Seizures Ended During Stim | 61.3 | 41.7 | 0 | 83.3 | 75.0 | 50.0

6. Secondary Outcome: Assesses Changes in Seizure Severity Based on Physician Reported Questionnaire (NHS3)
Description: Investigators completed the National Hospital Seizure Severity Scale (NHS3) questionnaire at screening, at the end of the EMU stay (provided a seizure occurred during the EMU stay), and at follow-up visits. Severity was evaluated by seizure type. The range of NHS3 scale is 1-27 with 1 being the least severe and 27 being the most severe.
  Negative median value means improvement.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Median (Full Range); unit: units on a scale
Groups:
- Complex Partial Seizure (CPS); CPS w/2nd GTC; Simple Partial Seizure (SPS): NHS3 Scores at Follow-Up Visits
Arm/Group | Complex Partial Seizure (CPS) | CPS w/2nd GTC | Simple Partial Seizure (SPS)
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Baseline to 3 Months; n=17,2,9 | -2.0 [-9.5 to 2.0] | -3.5 [-4.0 to -3.0] | 0.0 [-2.0 to 3.0]
  Baseline to 6 Months; n=17,4,11 | -0.5 [-12.0 to 3.0] | -1.0 [-9.0 to 2.0] | 0.0 [-2.0 to 1.0]
  Baseline to 12 Months; n=18,6,10 | -1.0 [-12.0 to 3.0] | -3.0 [-7.0 to 3.0] | 0.0 [-2.0 to 2.0]
  Baseline to 18 Months; n=15, 6, 9 | -3.0 [-5.0 to 4.0] | -2.5 [-6.0 to -1.0] | 0.0 [-6.0 to 10.0]
Statistical Analysis 1: Comparison: Complex Partial Seizure (CPS); Baseline to 3 months; Test type: Superiority or Other; p = 0.008, Signed Rank Test; Null hypothesis: change from the baseline is equal to zero. The alternative hypothesis: change from the baseline is not equal to zero
Statistical Analysis 2: Comparison: Complex Partial Seizure (CPS); Baseline to 6 months; Test type: Superiority or Other; p = 0.040, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Complex Partial Seizure (CPS); Baseline to 12 months; Test type: Superiority or Other; p = 0.033, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: CPS w/2nd GTC; Baseline to 3 months; Test type: Superiority or Other; p = 0.500, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: CPS w/2nd GTC; Baseline to 6 months; Test type: Superiority or Other; p = 0.750, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: CPS w/2nd GTC; Baseline to 12 months; Test type: Superiority or Other; p = 0.156, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Simple Partial Seizure (SPS); Baseline to 3 months; Test type: Superiority or Other; p = 0.938, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Simple Partial Seizure (SPS); Baseline to 6 months; Test type: Superiority or Other; p = 0.250, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Simple Partial Seizure (SPS); Baseline to 12 months; Test type: Superiority or Other; p = 0.999, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 10: Comparison: Complex Partial Seizure (CPS); Baseline to 18 Months; Test type: Superiority or Other; p = 0.057, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 11: Comparison: CPS w/2nd GTC; Baseline to 18 Months; Test type: Superiority or Other; p = 0.031, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 12: Comparison: Simple Partial Seizure (SPS); Baseline to 18 Months; Test type: Superiority or Other; p = 0.625, Signed Rank Test; [statistical method as in outcome 6, analysis 1]

7. Secondary Outcome: Assess Changes in Seizures Severity, Intensity & Post-Ictal Recovery Based on Patient Completed Questionnaire (SSQ)
Description: Clinical outcomes such as seizure severity, intensity and post-ictal duration were also assessed during the long-term follow-up visits (3, 6, 12, 18 months) with patient reported questionnaires (SSQ; Seizure Severity Questionnaire). The range for SSQ (all sub-scores) is 1-7 with 1 being the least severe and 7 being the most severe.
  Mean SSQ scores at 3, 6, 12 and 18 months were compared to baseline. A change from baseline is calculated as baseline minus follow-up visit score to correspond to the Minimally Important Change (MIC) criteria as defined in the Scoring Scheme for SSQ v2. Questionnaire.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- SSQ Scores at 3 Months; SSQ Scores at 6 Months; SSQ Scores at 12 Months; SSQ Scores at 18 Months: Change From Baseline at Each Category
Arm/Group | SSQ Scores at 3 Months | SSQ Scores at 6 Months | SSQ Scores at 12 Months | SSQ Scores at 18 Months
Number analyzed (Participants) | 20 | 20 | 20 | 20
Units on a Scale
  SSQ Total Score n=19,20,20,17 MIC=0.48 | 1.349 (1.488) | 1.442 (1.736) | 1.469 (1.908) | 1.711 (1.389)
  Activity During Seizure; n=15,17,16, 15 MIC=0.5 | 1.567 (2.890) | 1.294 (2.840) | 1.469 (2.895) | 1.200 (2.242)
  Overall Recovery; n=19,20,19,17 MIC=0.39 | 1.298 (2.215) | 1.489 (2.570) | 1.942 (2.817) | 1.922 (1.862)
  Overall Severity; n=19,20,20,17 MIC=0.48 | 1.246 (2.137) | 1.383 (2.238) | 1.767 (2.717) | 1.765 (1.711)
  Postictal Emotional Recovery n=19,20,19,17MIC=0.34 | 1.351 (2.430) | 1.733 (2.494) | 1.825 (2.838) | 1.922 (2.631)
  Postictal Physical Recovery; n=19,20,19,17MIC=0.48 | 1.123 (2.803) | 1.450 (3.789) | 2.088 (3.778) | 2.098 (2.710)
  Postictal Cognitive Recovery;n=19,20,19,17MIC=0.42 | 1.421 (3.166) | 1.283 (3.436) | 1.912 (3.878) | 1.745 (2.917)
Statistical Analysis 1: Comparison: SSQ Scores at 3 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.0008, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: SSQ Scores at 3 Months; Activity During Seizure Score; Test type: Superiority or Other; p = 0.0544, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: SSQ Scores at 3 Months; Overall Recovery Score; Test type: Superiority or Other; p = 0.0207, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: SSQ Scores at 3 Months; Overall Severity Score; Test type: Superiority or Other; p = 0.0163, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: SSQ Scores at 3 Months; Postictal Emotional Recovery Score; Test type: Superiority or Other; p = 0.0156, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: SSQ Scores at 3 Months; Postictal Physical Recovery Score; Test type: Superiority or Other; p = 0.0742, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: SSQ Scores at 3 Months; Postictal Cognitive Recovery Score; Test type: Superiority or Other; p = 0.0884, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: SSQ Scores at 6 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.0007, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: SSQ Scores at 6 Months; Activity During Seizure; Test type: Superiority or Other; p = 0.1173, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 10: Comparison: SSQ Scores at 6 Months; Overall Recovery; Test type: Superiority or Other; p = 0.0214, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 11: Comparison: SSQ Scores at 6 Months; Overall Severity; Test type: Superiority or Other; p = 0.0114, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 12: Comparison: SSQ Scores at 6 Months; Postictal Emotional Recovery; Test type: Superiority or Other; p = 0.0078, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 13: Comparison: SSQ Scores at 6 Months; Postictal Physical Recovery; Test type: Superiority or Other; p = 0.0875, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 14: Comparison: SSQ Scores at 6 Months; Postictal Cognitive Recovery; Test type: Superiority or Other; p = 0.1526, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 15: Comparison: SSQ Scores at 12 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.0031, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 16: Comparison: SSQ Scores at 12 Months; Activity During Seizure; Test type: Superiority or Other; p = 0.0828, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 17: Comparison: SSQ Scores at 12 Months; Overall Recovery; Test type: Superiority or Other; p = 0.0092, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 18: Comparison: SSQ Scores at 12 Months; Overall Severity; Test type: Superiority or Other; p = 0.0096, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 19: Comparison: SSQ Scores at 12 Months; Postictal Emotional Recovery; Test type: Superiority or Other; p = 0.0234, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 20: Comparison: SSQ Scores at 12 Months; Postictal Physical Recovery; Test type: Superiority or Other; p = 0.0284, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 21: Comparison: SSQ Scores at 12 Months; Postictal Cognitive Recovery; Test type: Superiority or Other; p = 0.0679, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 22: Comparison: SSQ Scores at 18 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.0003, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 23: Comparison: SSQ Scores at 18 Months; Activity During Seizures Score; Test type: Superiority or Other; p = 0.0728, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 24: Comparison: SSQ Scores at 18 Months; Overall Recovery Score; Test type: Superiority or Other; p = 0.0005, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 25: Comparison: SSQ Scores at 18 Months; Overall Severity Score; Test type: Superiority or Other; p = 0.0005, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 26: Comparison: SSQ Scores at 18 Months; Postictal Emotional Recovery Score; Test type: Superiority or Other; p = 0.0078, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 27: Comparison: SSQ Scores at 18 Months; Postictal Physical Recovery Score; Test type: Superiority or Other; p = 0.0078, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 28: Comparison: SSQ Scores at 18 Months; Postictal Cognitive Recovery Score; Test type: Superiority or Other; p = 0.0273, Signed Rank Test; [statistical method as in outcome 6, analysis 1]

8. Secondary Outcome: Assess Changes From Baseline in Quality of Life Based on Patient Completed Questionnaire (QOLIE-31-P)
Description: Adult subjects (18 years and older) completed the Quality of Life in Epilepsy-Patient-Weighted (QOLIE-31-P) survey questionnaire at screening and safety follow-up visits. The range for QOLIE-31-P (Sub-domains) scale is 0-100. The higher the score the better quality of life.
  Mean QOLIE-31-P scores at 3, 6, 12 and 18 months were compared to baseline. MIC Thresholds as defined in Simon Borghs, Christine de la Loge, Joyce A. Cramer, defining minimally important change in QOLIE-31-P scores.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- QOLIE-31-P Scores at 3-Months; QOLIE-31-P Scores at 6-Months; QOLIE-31-P Scores at 12-Months; QOLIE-31-P Scores at 18-Months: Change From Baseline at Each Category
Arm/Group | QOLIE-31-P Scores at 3-Months | QOLIE-31-P Scores at 6-Months | QOLIE-31-P Scores at 12-Months | QOLIE-31-P Scores at 18-Months
Number analyzed (Participants) | 20 | 20 | 20 | 20
Units on a Scale
  QOLIE Overall Total Score; n=20,20,19,18 MIC=5.19 | 11.0 (18.8) | 11.8 (19.1) | 13.3 (23.6) | 14.4 (24.1)
  Energy/Fatigue; n=20,20,20,19 MIC=5.25 | 2.7 (25.6) | 4.0 (22.7) | 8.8 (26.1) | 6.1 (32.4)
  Emotional well being; n=20,20,20,18 MIC=4.76 | 7.7 (25.4) | 8.7 (27.7) | 10.1 (33.5) | 3.0 (36.5)
  Social Functioning; n=19,20,20,18 MIC=3.95 | 11.0 (25.9) | 11.0 (18.2) | 9.6 (25.6) | 12.5 (30.1)
  Cognitive Functioning; n=20,20,20,19 MIC=5.34 | 19.2 (24.6) | 19.0 (24.4) | 16.6 (30.4) | 16.3 (32.7)
  Medication Effects; n=19,20,19,19 MIC=5.0 | 10.3 (33.1) | 8.1 (30.0) | 10.4 (37.5) | 16.7 (33.2)
  Seizure Worry; n=20,20,20,19 MIC=7.42 | 16.4 (32.2) | 16.9 (28.6) | 20.9 (27.6) | 23.3 (29.2)
  Overall Quality of Life; n=20,20,19,17 MIC=6.42 | 10.6 (24.7) | 14.6 (27.8) | 13.1 (30.6) | 19.1 (29.5)
Statistical Analysis 1: Comparison: QOLIE-31-P Scores at 3-Months; QOLIE Overall Total; Test type: Superiority or Other; p = 0.0192, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: QOLIE-31-P Scores at 3-Months; Energy/Fatigue; Test type: Superiority or Other; p = 0.8069, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: QOLIE-31-P Scores at 3-Months; Emotional well being; Test type: Superiority or Other; p = 0.2416, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: QOLIE-31-P Scores at 3-Months; Social Functioning; Test type: Superiority or Other; p = 0.1111, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: QOLIE-31-P Scores at 3-Months; Cognitive Functioning; Test type: Superiority or Other; p = 0.0014, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: QOLIE-31-P Scores at 3-Months; Medication Effects; Test type: Superiority or Other; p = 0.3247, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: QOLIE-31-P Scores at 3-Months; Seizure Worry; Test type: Superiority or Other; p = 0.0826, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: QOLIE-31-P Scores at 3-Months; Overall Quality of Life; Test type: Superiority or Other; p = 0.1040, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: QOLIE-31-P Scores at 6-Months; QOLIE Overall Total; Test type: Superiority or Other; p = 0.0094, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 10: Comparison: QOLIE-31-P Scores at 6-Months; Energy/Fatigue; Test type: Superiority or Other; p = 0.5874, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 11: Comparison: QOLIE-31-P Scores at 6-Months; Emotional well being; Test type: Superiority or Other; p = 0.1508, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 12: Comparison: QOLIE-31-P Scores at 6-Months; Social Functioning; Test type: Superiority or Other; p = 0.0136, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 13: Comparison: QOLIE-31-P Scores at 6-Months; Cognitive Functioning; Test type: Superiority or Other; p = 0.0015, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 14: Comparison: QOLIE-31-P Scores at 6-Months; Medication Effects; Test type: Superiority or Other; p = 0.3522, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 15: Comparison: QOLIE-31-P Scores at 6-Months; Seizure Worry; Test type: Superiority or Other; p = 0.0240, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 16: Comparison: QOLIE-31-P Scores at 6-Months; Overall Quality of Life; Test type: Superiority or Other; p = 0.0353, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 17: Comparison: QOLIE-31-P Scores at 12-Months; QOLIE Overall Total Score; Test type: Superiority or Other; p = 0.0361, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 18: Comparison: QOLIE-31-P Scores at 12-Months; Energy/Fatigue; Test type: Superiority or Other; p = 0.1921, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 19: Comparison: QOLIE-31-P Scores at 12-Months; Emotional well being; Test type: Superiority or Other; p = 0.1639, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 20: Comparison: QOLIE-31-P Scores at 12-Months; Social Functioning; Test type: Superiority or Other; p = 0.1738, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 21: Comparison: QOLIE-31-P Scores at 12-Months; Cognitive Functioning; Test type: Superiority or Other; p = 0.0401, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 22: Comparison: QOLIE-31-P Scores at 12-Months; Medication Effects; Test type: Superiority or Other; p = 0.2753, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 23: Comparison: QOLIE-31-P Scores at 12-Months; Seizure Worry; Test type: Superiority or Other; p = 0.0056, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 24: Comparison: QOLIE-31-P Scores at 12-Months; Overall Quality of Life; Test type: Superiority or Other; p = 0.1173, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 25: Comparison: QOLIE-31-P Scores at 18-Months; QOLIE Overall Total; Test type: Superiority or Other; p = 0.0268, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 26: Comparison: QOLIE-31-P Scores at 18-Months; Energy/Fatigue Final; Test type: Superiority or Other; p = 0.4406, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 27: Comparison: QOLIE-31-P Scores at 18-Months; Emotional Well Being Final; Test type: Superiority or Other; p = 0.7926, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 28: Comparison: QOLIE-31-P Scores at 18-Months; Social Functioning Final; Test type: Superiority or Other; p = 0.0987, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 29: Comparison: QOLIE-31-P Scores at 18-Months; Cognitive Functioning Final; Test type: Superiority or Other; p = 0.0361, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 30: Comparison: QOLIE-31-P Scores at 18-Months; Medication Effects Final; Test type: Superiority or Other; p = 0.0615, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 31: Comparison: QOLIE-31-P Scores at 18-Months; Seizure Worry; Test type: Superiority or Other; p = 0.0024, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 32: Comparison: QOLIE-31-P Scores at 18-Months; Overall Quality of Life; Test type: Superiority or Other; p = 0.0155, Signed Rank Test; [statistical method as in outcome 6, analysis 1]

9. Secondary Outcome: Assess Changes From Baseline in Seizure Frequency
Description: Seizure frequency was calculated at 3, 6,12 and 18 month follow-up visits based on seizure diary information and compared to baseline estimates. Response rate was computed and summarized for partial seizures (SPS, CPS and CPS with 2nd GTCs) and overall seizure types as the proportion of patients that achieved ≥50% seizure reduction per month from baseline by visit.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Partial Onset Seizure Responder Rate: Partial Onset Seizures (SPS, CPS, CPS with Secondary GTC)
- Overall Seizure Responder Rate: Overall Seizure (All Seizure Types)
Arm/Group | Partial Onset Seizure Responder Rate | Overall Seizure Responder Rate
Number analyzed (Participants) | 20 | 20
Percentage of Participants
  At 3-Month Visit; n=5,4 | 25 [8.66 to 49.10] | 20 [5.73 to 43.66]
  At 6-Month Visit; n=7,7 | 35 [15.39 to 59.22] | 35 [15.39 to 59.22]
  At 12-Month Visit; n=10,10 | 50 [27.20 to 72.80] | 50 [27.20 to 72.80]
  At 18-Month Visit; n=11,11 | 55 [31.53 to 76.94] | 55 [31.53 to 76.94]

10. Secondary Outcome: Assess Percent Changes in Antiepileptic Drug (AED) Load From Baseline
Description: AED load were collected and measured from baseline.The AED load is calculated as the sum of all ratios of the total daily dose of each medication taken on the day of the visit over the defined daily dose of the medication for the main indication according to the WHO database.
  Positive median value indicates increased drug load.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Median (Full Range); unit: Percent Change
Groups:
- AED Load: Percent Change From Baseline by Visit
Arm/Group | AED Load
Number analyzed (Participants) | 20
Percent Change
  At 3 months | 0 [0.00 to 30.00]
  At 6 months | 0 [-24.96 to 30.00]
  At 12 months | 3.35 [-59.55 to 52.74]
  At 18 Months | 0 [-59.55 to 42.00]
Statistical Analysis 1: Comparison: AED Load; 3 months; Test type: Superiority or Other; p = 0.0625, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: AED Load; 6 months; Test type: Superiority or Other; p = 0.1094, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: AED Load; 12 months; Test type: Superiority or Other; p = 0.0342, Signed Rank Test; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: AED Load; 18 Months; Test type: Superiority or Other; p = 0.5417, Signed Rank Test; [statistical method as in outcome 6, analysis 1]

11. Primary Outcome: Estimate the Effect Size Associated With Objective Measures and Patient Self-reports of Clinical Outcomes Including Seizure Frequency, Seizure Severity, Seizure Duration, Seizure Intensity, and Post-ictal Duration.
Description: The purpose for determining the effect size was to power a stage 2 study. At the conclusion of stage 1 of the E-37 study, it was determined that another study would not be necessary as it would not provide incremental clinical benefit information above what has already been collected. Therefore, computation of effect size was not necessary.
Time Frame: Up to 18 Month Visit-End of Study
Groups:
- VNS Therapy: ITT Population
Arm/Group | VNS Therapy
Number analyzed (Participants) | 0

12. Secondary Outcome: Assess All Adverse Events to Outline the Tolerability Profile of the AspireSR® VNS Therapy® System
Description: All adverse events (AEs) occurring during the study were collected and incidence rates tabulated by System Organ Class and Preferred Term utilizing MedDRA version 16.1 dictionary. The incidence profile was used to assess differences in near term tolerability rates relative to standard VNS Therapy.
Time Frame: From initial titration visit (approximately 2 weeks after implantation) up to End of Study
Population: ITT Population
Measure: Number; unit: Number of Participants
Groups:
- Number of Subjects: Experienced Adverse Events Greater Than 5% Incidence
Arm/Group | Number of Subjects
Number analyzed (Participants) | 20
Number of Participants
  Convulsion | 6
  Dysphonia | 6
  Oropharyngeal Pain | 3
  Stress | 3
  Urinary Tract Infection | 2
  Contusion | 2
  Dysphagia | 2
  Headache | 2
  Tooth Fracture | 2
  Umblical Hernia | 2

13. Secondary Outcome: Evaluation of Human Factors and Usability of the AspireSR® VNS Therapy® System.
Description: Usability survey data were collected from all site personnel who used the handheld programmer to evaluate the usability of the AspireSR® VNS Therapy® System.The device usability survey contained 17 questions that measure usability on a five-point Likert scale ranging from "Extremely Difficult" (5) to "Extremely Easy" (1). Site personnel were asked to assess usability of the software features, instructions for use, training materials, and overall usability of the system at four different time points. The time points include implant/recovery, the first day of EMU, the end of EMU, and the 6 month follow-up visit.
  Overall Usability was calculated as percentage of the users who found the overall usability of system to be "easy-2" or extremely easy-1".
Time Frame: Up to 6 Month Visit
Population: ITT Population
Measure: Number; unit: Percentage of Participants Rated 1 or 2
Groups:
- Implant/Recovery; EMU Day-1; EMU Discharge; 6-Month Visit: Users' Overall Assessment of Device Usability
Arm/Group | Implant/Recovery | EMU Day-1 | EMU Discharge | 6-Month Visit
Number analyzed (Participants) | 18 | 18 | 20 | 18
Percentage of Participants Rated 1 or 2 | 89 | 83 | 95 | 100

14. Secondary Outcome: Assess Changes in Healthcare Utilization: Inpatient Hospital Visits, Emergency Room Visits, Outpatient Hospitalizations and Physician Office Visits.
Description: At baseline and each follow-up visit, subjects completed a healthcare utilization questionnaire to report the number of unplanned inpatient hospitalizations, emergency room visits, outpatient hospitalizations, physician office visits.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Median (Full Range); unit: Visits
Groups:
- 3-Month; 6-Month; 12-Month; 18-Month: Since Last Visit Assessment
Arm/Group | 3-Month | 6-Month | 12-Month | 18-Month
Number analyzed (Participants) | 20 | 20 | 20 | 20
Visits
  Inpatient Hospital visits, n=20, 20, 20, 20 | 0 [0.00 to 0.00] | 0 [0.00 to 1.00] | 0 [0.00 to 1.00] | 0 [0.00 to 1.00]
  Emergency Room Visits, n=20, 20, 20, 20 | 0 [0.00 to 1.00] | 0 [0.00 to 2.00] | 0 [0.00 to 4.00] | 0 [0.00 to 2.00]
  Outpatient Hospital Visits, n=20, 20, 20, 19 | 0 [0.00 to 1.00] | 0 [0.00 to 1.00] | 0 [0.00 to 3.00] | 0 [0.00 to 1.00]
  Physician Office Visits, n=20, 20, 20, 20 | 0 [0.00 to 4.00] | 0 [0.00 to 4.00] | 0 [0.00 to 4.00] | 0 [0.00 to 8.00]

15. Secondary Outcome: Assess Changes in Healthcare Utilization: Number of Nights Spent at the Hospital
Description: At baseline and each follow-up visit, subjects completed a healthcare utilization questionnaire to report the number of nights spent at the hospital.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Median (Full Range); unit: Nights
Arm/Group | 3-Month | 6-Month | 12-Month | 18-Month
Number analyzed (Participants) | 20 | 20 | 20 | 20
Nights | 0 [0.00 to 0.00] | 0 [0.00 to 1.00] | 0 [0.00 to 1.00] | 0 [0.00 to 3.00]

16. Secondary Outcome: Assess Changes in Healthcare Utilization: Days Per Week Patients and Caregivers Could Not Work
Description: At baseline and each follow-up visit, subjects completed a healthcare utilization questionnaire to report the number of days per week of missed work because of health reasons.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Median (Full Range); unit: Days Per Week
Arm/Group | 3-Month | 6-Month | 12-Month | 18-Month
Number analyzed (Participants) | 20 | 20 | 20 | 20
Days Per Week
  #of DD/WK Could not work or Play(Pt),n=18,18,19,20 | 0 [0.00 to 3.00] | 0 [0.00 to 7.00] | 0 [0.00 to 3.00] | 0 [0.00 to 7.00]
  #of DD/WK Could not Work(Caregiver),n=18, 20,17,15 | 0 [0.00 to 7.00] | 0 [0.00 to 7.00] | 0 [0.00 to 7.00] | 0 [0.00 to 7.00]

17. Secondary Outcome: Assess Changes in Healthcare Utilization: Number of Hours Per Week Caregivers Spent Caring for Patients.
Description: At baseline and each follow-up visit, subjects completed a healthcare utilization questionnaire to report the number of hours per week caregivers spent caring for patients.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Median (Full Range); unit: Hours Per Week
Arm/Group | 3-Month | 6-Month | 12-Month | 18-Month
Number analyzed (Participants) | 19 | 20 | 17 | 15
Hours Per Week | 2.0 [0.00 to 100.00] | 1.0 [0.00 to 56.00] | 4.0 [0.00 to 168.00] | 2.0 [0.00 to 168.00]

18. Secondary Outcome: Assess Changes in Healthcare Utilization: Number of Phone Calls to Physician
Description: At baseline and each follow-up visit, subjects completed a healthcare utilization questionnaire to report the number of phone calls to physicians.
Time Frame: Up to 18 Month Visit-End of Study
Population: ITT Population
Measure: Median (Full Range); unit: Phone Calls
Arm/Group | 3-Month | 6-Month | 12-Month | 18-Month
Number analyzed (Participants) | 20 | 20 | 20 | 19
Phone Calls | 0 [0.00 to 5.00] | 0 [0.00 to 3.00] | 0 [0.00 to 7.00] | 0 [0.00 to 10.00]

ADVERSE EVENTS:
Time Frame: After Implantation up to 18 months-End of Study
Groups:
- VNS Therapy - Safety Population: All adverse events were collected from baseline up to the end of study for all subjects treated/implanted with the AspireSR® VNS Therapy® system. Only the most common AEs (> 5%) are reported in the AE data table.
Arm/Group | VNS Therapy - Safety Population
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VNS Therapy - Safety Population (N=20)
Incision wound cellulitis (Surgical and medical procedures) | 1
Post-procedural hematoma (Surgical and medical procedures) | 1
Altered State of Consciousness (Nervous system disorders) | 1
Subdural Hematoma (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VNS Therapy - Safety Population (N=20)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 — 1 Related to Implantation Procedure, 5 Related to VNS Therapy Stimulation, 1 Related to Both VNS Therapy Stimulation and Implantation Procedure
Convulsion (Nervous system disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 — 2 Related to VNS Therapy Stimulation
Stress (Psychiatric disorders) | 3
Urinary Tract Infection (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 2 — 1 Reported to VNS Therapy Stimulation
Procedural Pain (Injury, poisoning and procedural complications) | 2 — All Related to Implantation Procedure
Tooth Fracture (Injury, poisoning and procedural complications) | 2
Vomiting (Gastrointestinal disorders) | 2 — 1 Related to VNS Therapy Stimulation
Dysphagia (Gastrointestinal disorders) | 2 — Related to VNS Therapy Stimulation
Headache (Nervous system disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Umblical Hernia (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
The small sample size and the absence of randomization did not allow conclusions about whether the AutoStim alone, or the combination of AutoStim and traditional VNS therapy modes, or some other factor was a cause of the observed beneficial effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted for sponsor's review if such publication contains Confidential Information or will adversely affect any intellectual property or proprietary right of the sponsor. The sponsor can require changes to the communication, but cannot extend the embargo set forth in the study agreement.